CLINICAL TRIAL: NCT01828541
Title: A Randomized Controlled Trial of Hypnosis for Pain and Itch Following Burn Injuries
Brief Title: Hypnosis for Pain and Itch Following Burn Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Shelley A. Wiechman, Associate Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000542
Record Dates: First submitted 2013-03-29; First posted 2013-04-10 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Burns
Keywords: Burn injuries
MeSH Terms: conditions — Burns | interventions — Hypnosis; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Other): Subjects in this condition will receive our standard care for itch, which includes a stepped based algorithm of medications.
  Interventions: Other: Standard of Care
- Hypnosis Condition (Experimental): Subjects in this condition will receive standard care plus the addition of 4 sessions of hypnosis delivered over a two month period.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — Patients in this group will receive standard care plus 4 sessions of hypnosis.
  Arms: Hypnosis Condition
Other: Standard of Care
  Arms: Standard Care

SUMMARY:
The purpose of this study is to determine whether hypnosis will decrease the intensity of either pain or itch in patients who have sustained a burn injury. Primary hypothesis: Hypnosis will provide more effective relief from post-burn itch and pain than a control intervention at 1-month, 3-months, 6-months and 1-year post-burn injury.

Secondary hypothesis 1: Subjects treated with hypnosis will report better sleep quality and fewer symptoms of Post Traumatic Stress Disorder (PTSD).

Secondary Hypothesis 2: Subjects treated with hypnosis will require less escalation of the gabapentin doses and have lower average pain scores than those in the control group.

Exploratory Hypothesis: Subjects who will randomize to the hypnosis treatment group early after injury will report lower rates of neuropathic pain and itch than subjects who will be enrolled in the study and receive hypnosis later in the healing process.

DETAILED DESCRIPTION:
This is a randomized, controlled study comparing two groups of subjects, those in the control (standard care) group and those in the experimental group (hypnosis).

Control subjects will receive treatment as usual, which consists of a standardized protocol for treating post-burn itch. This protocol is based on past research and combines medications in a stepped approach that establishes therapeutic decisions based on clearly defined criteria.

Subjects randomized to the experimental group will undergo four sessions of live hypnosis completed over a two month period. They will be provided with a Compact Disk (CD) of each session and instructed to listen to it daily. Post-hypnotic suggestions will address uncomfortable sensations, with additional suggestions for improved sleep and well-being. Subjects may be inpatient or outpatients.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Ability to provide informed consent for study participation
* ability to read and understand English
* Undergoing pharmacologic therapy for burn related itch according to the standard itch protocol
* Scoring of 4 out of 10 on the Numerical Rating Scale for average itch or pain

Exclusion Criteria:

* Age less than 18 or greater than 65
* Inability to provide informed consent
* Inability to read or understand English
* Delirium
* History of mania, paranoia, dissociation and current suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale for Average Itch | 48 hours, 1-, 3-, 6-, 12- months post-randomization
  Subjects will be asked to rate their average itch intensity over the previous 24-hour period using the 0 (no itch) to 10 (worst itch imaginable) scale. Change in this measures over time will be assessed.

SECONDARY OUTCOMES:
Change in Numerical Rating Scale for Pain | 48 hours, 1-. 3-. 6-, 12-months post-randomization
  Subjects will be asked to rate their average pain intensity over the past 24 hours using the 0(no pain) to 10 (worst pain imaginable) scale. Change in this measure over time will be assessed.
Change in Medical Outcomes Study of Sleep | 1-, 3-, 6-, 12-months post-randomization
  This tool measures six different sleep constructs. We will use the 9-item sleep problem index score. Change in this measure over time will be assessed.
Change in Leeds Assessment of Neuropathic Symptoms and Signs-Self report | 1-, 3-, 6-, 12-months post randomization
  A self report scale that is aimed at identifying neuropathic pain without the need for clinical examination. Change in this measure over time will be assessed.
Change in 5-D Itch Scale | 1-, 3-, 6-, 12 months post randomization
  Addresses the impact of itch over the previous two week period of time. Change in this measure over time will be assessed.
Change in Post-Traumatic Stress Disorder Checklist-Civilian version | 1-, 3-, 6-, 12-month post-randomization
  A 17-item scale that measures each of the Diagnostic and Diagnostic and Statistical Manual-IV (DSM-IV) symptoms of Post Traumatic Stress Disorder (PTSD). Change in this measure over time will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided